CLINICAL TRIAL: NCT02922218
Title: Prospective Multi-Centre Study of Prognostic Factors in Metastatic Castration-Resistant Prostate Cancer Patients Treated With Enzalutamide.
Brief Title: PROSENZA: Prospective Multi-Centre Study of Prognostic Factors in mCRPC Patients Treated With Enzalutamide.
Acronym: PROSENZA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Collaborators: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: IBIMA-CNIO-CP-01-2016; CNI-ENZ-2016-01 (Other: CNIO)
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Advanced Prostate Cancer; Castration Resistant; Enzalutamide
Keywords: metastatic Castration Resistant Prostate Cancer; Enzalutamide; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and archival FFPE
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enzalutamide: Enzalutamide 160 mg/day c/24h

SUMMARY:
PROSENZA is a prospective multicentre observational study in metastatic Castration-Resistant Prostate Cancer (mCRPC), designed to explore prognostic biomarkers in patients undergoing treatment with enzalutamide

DETAILED DESCRIPTION:
This study is a prospective biomarker study of patients with mCRPC undergoing treatment with enzalutamide as standard of care treatment. The participants will undergo serial pre- and post-therapy blood collection for biomarker analysis as part of the primary objective of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male age ≥ 18 years
2. Histologically confirmed adenocarcinoma of the prostate
3. ECOG Performance Status ≤ 2
4. Castration resistance must be documented with surgical or medical castration with serum testosterone < 50 ng/mL (< 2.0 nM).
5. Men diagnosed with at least one metastatic lesion on CT or bone scan.
6. Documented biochemical and/or radiographic progression to previous treatment according to PCWG2 criteria.
7. Patients who are candidates for standard of care treatment with enzalutamide 160 mg every 24 hours.
8. Availability of formalin-fixed paraffin-embedded blocks from the prostate biopsy and/or radical prostatectomy.
9. Acceptable hematological, hepatic and renal functions.

Exclusion Criteria:

1. Previous cancer diagnosis, except those patients who had a localized malignant tumour and who are five years cancer-free or those diagnosed with skin cancers (of non-melanoma type) or excised in situ carcinomas.
2. Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic Castration-Resitant Prostate Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To assess the prognostic value for overall survival of androgen receptor splicing variant 7 (AR-V7) and/or AR amplification in mCRPC patients | Initially 48 months, currently 60 months

SECONDARY OUTCOMES:
To analyze the correlation between biochemical and/or radiological response with AR-V7 expression and/or AR amplification in mCRPC patients treated with Enzalutamide. | Initially 48 months, currently 60 months
To assess AR-V7 expression and/or AR amplification changes before and after enzalutamide treatment | Initially 48 months, currently 60 months
To explore the correlation between AR-V7 expression and AR amplification with other biomarkers as testosterone serum levels, PTEN loss or TMPRSS-ERG fusions in mCRPC patients treated with Enzalutamide | Initially 48 months, currently 60 months
To validate the prognostic value of classical nomograms designed to assess the outcomes of mCRPC patients in these patients | Initially 48 months, currently 60 months

OTHER OUTCOMES:
To validate the independent prognostic value of the gene-expression signature from peripheral blood described by Olmos et al (Lancet Oncol 2012) on overall survival of mCRPC patients | Initially 48 months, currently 60 months
To correlate the presence of somatic and/or germinal mutations with the outcomes of these patients | Initially 48 months, currently 60 months

CONTACTS AND LOCATIONS:
Overall Officials: David Olmos, MD, Study Chair — CNIO-Centro Nacionald e Investigaciones Oncológicas
Locations (26):
- Spain (26):
  - Hospital Arquitecto Marcide, Ferrol, A Coruña
  - Hospital Universitario de Santiago, Santiago de Compostela, A Coruña
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Althaia Manresa, Manresa, Barcelona
  - Hospital de Especialidades de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Costa del Sol, Marbella, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Fundacion Centro Oncologico de Galicia, A Coruña
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital de Burgos, Burgos
  - Hospital de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario Gregorio Maranon, Madrid
  - Coordination PROCURE-Centro Nacional de Investigaciones Oncologicas, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Regional Universitario Virgen de la Victoria, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Messeguer, Murcia
  - Hospital Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No